CLINICAL TRIAL: NCT05930587
Title: Effect of Lower Extremities Cold Immersion Applied to Patients With Varicose Veins on Quality of Life, Anxiety and Symptoms
Brief Title: Effect of Cold Immersion on Patients With Varicose Vein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nevra KALKAN, Res. Asst. PhD NEVRA KALKAN, Faculty of Nursing, Department of Surgical Nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziUNKalkan
Record Dates: First submitted 2023-06-13; First posted 2023-07-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Varicose Veins of Lower Limb

STUDY DESIGN:
Intervention Model Description: 2 groups (experimental group and control group)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients in the experimental and control groups in the study will be assigned to the groups by a statistician using a computer program, and the list of patients in the experimental and control groups will be submitted to the head nurse of the cardiovascular surgery clinic.Researchers will not be informed about which group the patients are in.
  In the research, the application of cold immersion to the patients in the experimental group will be explained by the nurse in charge, and data collection forms will be applied to both the experimental and control groups by the head nurse.
  As the patients will do the application directly themselves, blinding will not be possible.
  In addition, codes in the form of x and y will be given to the experimental and control groups and support will be received from another statistical expert.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold water immersion (Experimental): The experimental group will be informed about the lower extremity cold immersion bath during the outpatient clinic controls and will be given a liquid meter digital thermometer that will allow them to check the cold water temperature at home. Patients will then be asked to do the lower extremity cold water immersion bath every day in their own home, for a total of four weeks, lasting 20 minutes in the evening before going to sleep.
  It is recommended that the cold dip bath last for 20 minutes and the temperature of the water should be 15 0C for it to be effective on the symptoms.
  At the end of four weeks, patients will be informed that they should come to the outpatient clinic again. When the patients come to the outpatient clinic, information about the application will be repeated and data collection forms will be applied by face-to-face interview method.
  Interventions: Other: Cold water immersion
- Control (No Intervention): No intervention will be made to the control group, only the data will be collected at the same time as the study group.

INTERVENTIONS:
Other: Cold water immersion — Cold water immersion (15 degree celsius, 20 minutes)
  Arms: Cold water immersion

SUMMARY:
In the literature, it is stated that cold water immersion to lower extremities is effective on the symptoms of the disease. Studies have shown that cold water immersion, which is one of the cold application methods, has effects on increasing joint mobility, reducing pain, reducing stress, anxiety, depression, and increasing quality of life etc.

For this reason, the study is planned as a randomized controlled interventional study to determine the effect of cold water immersion directly to the lower extremity in the preoperative period of patients with varicose veins on quality of life, anxiety and symptoms experienced.

DETAILED DESCRIPTION:
The experimental group will be informed about the lower extremity cold immersion bath during the outpatient clinic controls and will be given a liquid meter digital thermometer that will allow them to check the cold water temperature at home. Patients will then be asked to do the lower extremity cold water immersion bath every day in their own home, for a total of four weeks, lasting 20 minutes in the evening before going to sleep.

It is recommended that the cold water immersion for 20 minutes and the temperature of the water should be 15 0C for it to be effective on the symptoms.

At the end of four weeks, patients will be informed that they should come to the outpatient clinic again. When the patients come to the outpatient clinic, information about the application will be repeated and data collection forms will be applied by face-to-face interview method.

To the patients in the control group; during the research process, routine outpatient controls will be made and no attempt will be made during the research.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65
* Those who have been diagnosed with lower extremity varicose disease for at least 1 year
* Those who have not had previous surgery due to varicose veins
* No visual, hearing and sensory impairment/neurosensor disorder problem
* No mental status disorder
* With intact skin integrity and no open wounds
* No circulatory disorder

Exclusion Criteria:

* The patient has a known cold allergy or hypersensitivity to cold
* Patient having surgery during the study
* The patient's desire to withdraw from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2023-10-25 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The Patient Questionnaire | four weeks
  This form was created by the researcher based on the literature. This form consists of questions which sociodemographic characteristics (age, gender, body mass index, marital status, living people, educational status, employment status, economic status), characteristics of health status (presence of chronic diseases, drugs used regularly, smoking and alcohol use), characteristics of varicose disease (how many years have varicose veins, which leg has varicose veins, family history of varicose veins, previous surgery for varicose veins and use of varicose stockings), and physical symptoms experienced due to varicose veins (expected to score according to 0-10 evaluation scale). according to the characteristics (how many years have varicose disease, which leg has varicose veins, family history of varicose veins, previous surgery for varicose veins and using varicose stockings).

SECONDARY OUTCOMES:
VEINES-QOL/Sym | four weeks
  VEINES-QOL/Sym is a standardised, 26-item, patient-reported questionnaire to assess the severity and frequency of venous insufficiency symptoms (questions 1,7; 10 items: heaviness, pain, leg swelling, night cramps, fatigue, burning sensation, throbbing sensation, itching, numbness in the legs, pain intensity), time of day when the symptoms are most pronounced (1 item, question 2), changes in the severity of symptoms during the past year (1 item, question 3), limitations in daily activities associated with venous insufficiency (9 item, questions 4,5,6), and the psychological impact on the functional status of patients with venous insufficiency measured during the previous 4 weeks (5 items, question 8). The scores are transformed as described in (14); the higher the result the better the quality of life.

OTHER OUTCOMES:
State and Trade Anxiety Inventory (STAI) | four weeks
  The STAI-X is an extensively used self-administered inventory of two sections containing 20 items each, designed to explore anxiety in its temporary condition of "state anxiety" (STAI-S) and the more general and longstanding quality of "trait anxiety" (STAI-T). The STAI-S assesses how respondents feel "right now, at this moment", and the STAI-T targets how respondents "generally feel". Each item is scored on a 4-point Likert scale, with choices ranging from 1 ("not at all") to 4 ("very much so") for the state scale, and 1 ("almost never") to 4 ("almost always") for the trait scale. The minimum score for each section is 20, with a maximum score of 80. A total score of 40 or more indicates an anxious condition. The higher the score is, the more severe the anxiety condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevra Kalkan, Ankara, Gazi University Faculty of Nursing, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- See also: Related Info — https://orcid.org/0000-0003-4536-7933